CLINICAL TRIAL: NCT04356170
Title: A Phase II Randomized Trial, Non Comparative, Evaluating Chemotherapy Associated Cisplatin, 5-fluorouracil and Docetaxel at Adapted Doses in Patients With Locally Advanced Squamous Cell Carcinoma
Brief Title: Trial Evaluating Adapted Chemotherapy in Patients With Squamous Carcinoma
Acronym: TPFmORL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Groupe Oncologie Radiotherapie Tete et Cou (Other)
Collaborators: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GORTEC 2019-01
Record Dates: First submitted 2020-04-10; First posted 2020-04-22 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Cancer of Head and Neck
Keywords: ORL cancer without front door, TPFm, inoperable tumor
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Docetaxel; Cisplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TPF (docetaxel, cisplatine, 5-FU) (Active Comparator): Docetaxel, cisplatine, 5-FU administered, every 3 weeks for a total of 3 cycles
  Interventions: Drug: Docetaxel; Drug: Cisplatin; Drug: Fluoro Uracil
- TPFm (docetaxel, cisplatine, 5-FU) modifié (Experimental): Docetaxel, cisplatine, 5-FU administered, every 2 weeks for a total of 6 cycles
  Interventions: Drug: Docetaxel; Drug: Cisplatin; Drug: Fluoro Uracil

INTERVENTIONS:
Drug: Docetaxel — Docetaxel 75 mg/m² administered at D1 of each cure, every 3 weeks by intravenous infusion in 1 hour
Drug: Cisplatin — cisplatine 75 mg/m² administered at D1 of each cure, every 3 weeks by intravenous infusion in 1 hour
Drug: Fluoro Uracil — 750 mg/m²/j administered continuously at D1 to D5 of each cure, every 3 weeks by intravenous infusion ( so 120 hours)

SUMMARY:
The objective of this study is to evaluate the efficacity of the combination of cisplatin-5-FU and docetaxel in adapted doses in term of response to treatment without toxicity

.

DETAILED DESCRIPTION:
After explaining the treatment modalities, having read and explained the information letter to them, patients who have signed the consent to participate in the trial and who meet the inclusion criteria will be enrolled and randomized in the trial .

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven squamous cell carcinoma of the head and neck from one or more of the following primary sites: oral cavity, oropharynx, hypopharynx or larynx, lymphadenopathy without front door
2. Inoperable tumor or tumor whose surgery would be multilating.

   The non-operability criteria are:
   * Technically impossible resection: fixation / invasion of the tumor at the base of the skull or at the cervical vertebrae, nasopharynx involved, lymph nodes
   * Medical selection based on low surgical curability. This category includes all T3-T4 and all N2-N3 (AJCC 8th edition, June 2018)
   * Medical selection based on an organ preservation strategy
3. Patient not previously treated for ORL cancer
4. Age > 18 and < 75 years
5. PS 0 or 1 according to WHO
6. At least one lesion measurable according to the RECIST 1.1 criteria
7. Patient who can receive TPF according to the following criteria:

   * Adequate hematological function: neutrophils ³ 1.5 x 109 / l, platelets *100 x 109 / l, hemoglobin 10 g / dl (or 6.2 mmol / l)
   * Adequate renal function: calculated creatinine clearance (Cockroft & Gault) or measured ³ 60 ml / min.
   * Adequate liver function: normal total bilirubin; ASAT and ALAT less than or equal to 1.5 ´ LNS; PAL less than or equal to 2.5 X LNS
   * Grade <2 peripheral neuropathy according to NCI CTCAE v5.0
   * No clinical impairment of hearing function
   * For patients aged 71 to 74, PS at 0 and considered non-geriatrically fragile (G8 questionnaire and multidimensional assessments proposed by the GERICO group (ADL, MMSE, GDS scale, nutrition, motor skills and balance, geographic and personal situation and assessments) thymic))
8. Estimated life expectancy greater than or equal to 3 months
9. Weight loss of less than 10% during the 3 months before randomization
10. Patient understanding French and able to complete quality of life questionnaires
11. Patient having given written consent before any specific protocol procedure
12. Affiliation to a social security scheme or beneficiary of such a scheme
13. Women of childbearing potential and sexually active men agreeing to use effective contraceptive methods for the duration of treatment and at least 6 months after the last administration of study treatments
14. Patient agrees not to donate sperm for the duration of the treatment and at least 6 months after the last administration of the study treatments
15. Absence of deficiency in dihydropyrimidine dehydrogenase activity determined by uracilemia assay (Uracilemia < 16 ng/mL)

Exclusion Criteria:

1. Cancers of the nasopharynx, sinuses or nasal cavities, and any histology other than squamous cell carcinoma
2. Vaccination against recent or planned yellow fever
3. Known deficiency in dihydropyrimidine dehydrogenase (DPD) or determined by the determination of uricemia.
4. History of other cancer except in situ cervical cancer or controlled basal cell carcinoma. Patients in remission from cancer treated more than 3 years ago are eligible. Patients treated by surgery alone for ORL cancer in the previous 3 years are eligible.
5. Previous treatment of an ORL cancer by chemotherapy or radiotherapy. Patients treated by surgery alone for ORL cancer in the previous 3 years are eligible).
6. Presence of distant metastasis.
7. Participation in a therapeutic trial in the 30 days preceding randomization
8. Concomitant anticancer treatment
9. Patient under chronic treatment (3 months) with corticosteroid whose daily dosage is 10 mg / day of methylprednisolone or equivalent
10. Other existing serious medical pathologies (non-exhaustive list):

    * Uncontrolled cardiac pathology despite adequate treatment
    * Myocardial infarction in the 6 months preceding randomization
    * Neurological or psychiatric history such as dementia, convulsions
    * Active infection
    * Significant gastrointestinal abnormalities, including those that require parenteral nutrition, active peptic ulcer, and history of surgeries affecting absorption
    * Obstructive pulmonary disease requiring hospitalization in the year preceding randomization
    * Uncontrolled type II diabetes or other corticosteroid contraindications.
    * Moderate or severe eczema
11. Known hypersensitivity to docetaxel, cisplatin 5FU or one of their excipients.
12. Intended concomitant use of phenytoin, carbamazepine, barbiturates or rifampicin
13. Presence, upon selection, of psychological, family, social or geographic factors likely to influence the patient's compliance with the study and monitoring protocol.
14. Pregnant or lactating woman
15. Patient (male or female) of reproductive age who is unable or unwilling to take adequate contraceptive measures during treatment and up to 6 months after the last treatment is administered.
16. Persons deprived of their liberty, under guardianship or curatorship

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2021-02-04 (Actual); Primary Completion 2025-08-05 (Actual); Study Completion 2025-08-05 (Actual)

PRIMARY OUTCOMES:
Efficacity of combination of TPFm | 8 weeks after the end of treatment
  Success rate of patients at 8 weeks

OTHER OUTCOMES:
Overall survival | 3 months after the end of treatment
  The time from date of randomization to date of death due to any cause
Progression free survival | 3 months after the end of treatment
  The time from date randomization to date of first evidence of progression
incidence of local and/or locorégional failure | 3 months after the end of treatment
Laryngeal preservation | 3 months after the end of treatment
incidence of distant metastatic failure | 3 months after the end of treatment
  The time from the date of randomization and the date of first evidence of metastatic progression, or the date of death, whatever the cause
Toxicities of complementary treatment to induction tretatment | 3 months after the end of treatment
  Rate of patients who received the whole of complementary treatment
QLQ-C30 questionnaires | 8 weeks, 6 months (3 months after the end of treatment) and 24 months after the end of treatment
  These questionnaires assess the impact of the desease and treatment on tthe patient's life
QLQ-H&N35 questionnaires | 8 weeks, 6 months (3 months after the end of treatment) and 24 months after the end of treatment
  These questionnaires assess the impact of the desease and treatment on tthe patient's life

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Leon Berard, Lyon, France